CLINICAL TRIAL: NCT02306811
Title: A Long-Term Follow-up Study Assessing the Safety and Efficacy of Vatelizumab in Multiple Sclerosis (MS) Patients Who Completed Treatment in Study DRI13839
Brief Title: Efficacy and Safety of Vatelizumab in Patients Who Completed Treatment in Study DRI13839
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study discontinued based on planned interim analysis of the primary endpoint. Not linked to any safety concern.
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LTS13840; 2014-003265-19 (EudraCT Number); U1111-1160-6120 (Other: UTN)
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Relapsing-remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vatelizumab Dose 1 (Experimental): Vatelizumab dose 1 every 4 weeks (Q4W) for 96 weeks
  Interventions: Drug: Vatelizumab
- Vatelizumab Dose 2 (Experimental): Vatelizumab dose 2 every 4 weeks (Q4W) for 96 weeks
  Interventions: Drug: Vatelizumab
- Vatelizumab Dose 3 (Experimental): Vatelizumab dose 3 every 4 weeks (Q4W) for 96 weeks
  Interventions: Drug: Vatelizumab
- Vatelizumab Dose 4 (Experimental): Vatelizumab dose 4 every 4 weeks (Q4W) for 96 weeks
  Interventions: Drug: Vatelizumab

INTERVENTIONS:
Drug: Vatelizumab — Pharmaceutical form:solution for infusion
  Route of administration: intravenous
  Other Names: SAR339658

SUMMARY:
Primary Objective:

To assess the long-term safety of vatelizumab in MS patients

Secondary Objective:

To assess the long-term efficacy of vatelizumab

DETAILED DESCRIPTION:
The maximum study duration per patient will be 192 weeks, including a Treatment Period of 96 weeks and Post-treatment Safety Follow-up Period of 96 weeks.

ELIGIBILITY:
Inclusion criteria:

Patients who completed the 12-week treatment period in DRI13839.

Exclusion criteria:

* Any clinically significant or ongoing adverse events, or laboratory abnormalities from DRI13839 that per Investigator judgment would adversely affect the patient's participation in the long-term extension study.
* Confirmed platelet count below the lower limit of normal at any time during DRI13839.
* Pregnancy or breast-feeding.
* Other protocol defined exclusion criteria may apply.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-02; Primary Completion 2016-04 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients experiencing adverse events | from Week 0 to Week 192

SECONDARY OUTCOMES:
Change in total volume of T2 lesions | from Week 0 to Week 84
Change in number of T1 hypointense lesions | from Week 0 to Week 84

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (18):
- United States (6):
  - Investigational Site Number 840004, Cullman, Alabama
  - Investigational Site Number 840005, Fort Collins, Colorado
  - Investigational Site Number 840007, Ormond Beach, Florida
  - Investigational Site Number 840001, Latham, New York
  - Investigational Site Number 840003, Round Rock, Texas
  - Investigational Site Number 840016, San Antonio, Texas
- Investigational Site Number 124001, Greenfield Park, Canada
- Poland (4):
  - Investigational Site Number 616001, Lodz
  - Investigational Site Number 616004, Lublin
  - Investigational Site Number 616003, Lublin
  - Investigational Site Number 616002, Szczecin
- Russia (7):
  - Investigational Site Number 643010, Kazan'
  - Investigational Site Number 643009, Moscow
  - Investigational Site Number 643006, Nizhny Novgorod
  - Investigational Site Number 643005, Nizhny Novgorod
  - Investigational Site Number 643008, Novosibirsk
  - Investigational Site Number 643002, Saint Petersburg
  - Investigational Site Number 643001, Saint Petersburg